CLINICAL TRIAL: NCT04403360
Title: Impact of the Erector Spinae Plane Block on the Postoperative Pain After Lumbar Spinal Stenosis Surgery: Single Blind Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block After Lumbar Spinal Stenosis Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinique Saint Pierre Ottignies (Other)
Responsible Party: Principal Investigator, Georges Samouri, Georges Samouri M.D., Clinique Saint Pierre Ottignies
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B707201837276
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Lumbar Spinal Stenosis; Erector Spinae Plane Block
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae plane Block (ESPB) group (Experimental): The ultrasound-guided ESPB was realized at T12 level (levo bupivacaine 0.25% + epinephrine 1:200.000 4mg.kg-1 body weight)after the induction of anesthesia but before the start of the surgery.
  Interventions: Procedure: ESPB
- Local anesthesia infiltration by the surgeon (Active Comparator): The surgeon infiltrates the surgical site after skin incision with local anesthetics (Levo Bupivacaïne 0.25% + epinephrine 1:200.000 4mg.kg-1 body weight)
  Interventions: Procedure: Local infiltration by the surgeon

INTERVENTIONS:
Procedure: ESPB — Ultrasound guided performance of ESPB at T12 level after the induction of anesthesia but before the start of the surgery
  Arms: Erector Spinae plane Block (ESPB) group
Procedure: Local infiltration by the surgeon — Local infiltration of anesthetics at surgical site after skin incision
  Arms: Local anesthesia infiltration by the surgeon

SUMMARY:
Lumbar spinae stenosis surgery is a frequent intervention resulting in important postoperative pain. Management of this postoperative pain is thus important. Different pain management therapies exist. The erector spinae plane (ESP) block was described in 2016. It involves the injection of local anesthetics into the interfascial plane, deep to erector spinae muscle, allowing the blockade of the dorsal and ventral rami of the thoracic spinal nerves. It was initially proposed for analgesia of costal fractures, pulmonary lobectomy and thoracic vertebrae. The ESP block (ESPB) could probably be extended to a large number of surgical procedures. ESPB has so far not been investigated in lumbar spinae stenosis surgery.

ELIGIBILITY:
Inclusion Criteria:

- Any lumbar spinae surgery on 2 or more lumbar levels

Exclusion Criteria:

* Contraindication to NSAID
* Allergy to any local anesthetics

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Total 24 h Piritramide consumption | 24 hours
  Total consumption of Piritramide consumption after surgery

SECONDARY OUTCOMES:
Quebec back pain disability scale (QBPDS) | At 2 months]
  A questionnaire developed to measure the level of functional disability for patients with low back pain

CONTACTS AND LOCATIONS:
Overall Officials: Georges SAMOURI, MD, Principal Investigator — Clinique Saint Pierre Ottignies
Locations (1):
- Clinique Saint Pierre, Ottignies, Brabant Wallon, Belgium

IPD SHARING:
Plan to Share IPD: No
All data will be presented in future manuscripts.

REFERENCES:
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016